CLINICAL TRIAL: NCT05932251
Title: Towards Precision Medicine for Diabetes in Pregnancy
Acronym: ToPMedDiP
Status: Suspended | Type: Observational
Why Stopped: Poor recruitment efficacy
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: NL80773.096.22
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes; Gestational Diabetes Mellitus
Keywords: insulin sensitivity; insulin secretion; continuous glucose monitoring; metformin; physical activity
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Motor Activity | interventions — Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low insulin sensitivity: Women will be classified as having low insulin sensitivity, if their Matsuda-index is in the lowest quartile of a reference cohort
  Interventions: Drug: Metformin
- Low insulin secretion: Women will be classified as having low insulin secretion if their Stumvoll-index is in the lowest quartile of a reference cohort
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — All patients are diagnosed with gestational diabetes and treated with metformin (per routine clinical practice

SUMMARY:
Rationale: Gestational diabetes is currently treated by the one-size-fits-all-approach. Treatment efficacy is poorly defined and inconsiderate of patients clinical presentation Objective: To characterize the efficacy of pharmacological treatment of gestational diabetes mellitus between patients with distinct metabolic phenotypes Study design: Prospective observational study, in metformin-treatment efficacy is compared between patients with GDM caused by insulin resistance and patients with GDM caused by low insulin secretion.

Study population: A prospective cohort of 103 women with diagnosed gestational diabetes mellitus treated by metformin.

Main study parameters/endpoints: Primary outcomes is the glucose-disposition-index in late pregnancy (35-37 weeks gestation) and requirement for supplemental insulin-treatment. Secondary outcomes include insulin sensitivity (Matsuda-index), insulin secretion (Stumvoll-index), HbA1c, gestational weight gain, body composition, physical activity, eating behavior, plasma biomarkers, glucose control, and maternal and infant pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* having a confirmed single, viable pregnancy past 20 weeks gestation.
* assigned to pharmacological (ie metformin) treatment for GDM.

Exclusion Criteria:

* pre-existing diabetes, hypertension (SBP >160 mmHg & DBP >110 mmHg)
* using medication related to study outcomes prior to GDM diagnosis (insulin, metformin, glyburide, systemic steroids, mood stabilizers, ADHD medication)
* smoking or using recreational drugs that may affect pregnancy outcomes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients, who are screened (selection per EXPECT-calculator risk for GDM >3.5% [26]) and diagnosed with GDM and treated with metformin are eligible. Per current clinical practice (IADPSG/WHO2013), GDM will be diagnosed at 24-28 weeks by a 75g-oral glucose-tolerance-test (OGTT), if plasma glucose concentrations are: fasting >5.1 mmol/L; 1-h >10 mmol/L; or 2-h >8.5 mmol/L.[2, 25] Metformin-treatment is initiated, if plasma glucose concentrations during the OGTT are: fasting >5.3 mmol/L; and postprandial: >7.8 mmol/L.
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
glucose-disposition-index | 35-37 weeks gestation
  glucose-disposition-index is calculated as product of Stumvoll- and Matsuda-index, assessed during a 75g-oral glucose tolerance test,

SECONDARY OUTCOMES:
Insulin treatment | 35-37 weeks gestation
  requirement for additional insulin treatment
HbA1c | 24-28 and 35-37 weeks gestation
  HbA1c concentration
Body weight | 24-28 and 35-37 weeks gestation
  Fasting body weight, kg
Body fat mass | 24-28 and 35-37 weeks gestation
  Fasting body fat mass, in kg
Physical Activity | 24-28 and 35-37 weeks gestation
  Average steps per day, measured over 7-day period using accelerometry
Dietary intake | 24-28 and 35-37 weeks gestation
  Average energy intake, measured over 7 days using online dietary records
Glucose control | 24-28 and 35-37 weeks gestation
  Time in range (3-10 mol/l), measured over 7 days using continuous glucose monitors
Delivery complications | Birth
  occurence and type of complications during delivery
Neonatal body weight | at birth, and at 6 weeks of age
  Neonatal body weight
Neonatal body length | at birth, and at 6 weeks of age
  Neonatal body length

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Most, PhD, Principal Investigator — Zuyderland Medisch Centrum; Jonas Ellerbrock, MD, PhDc, Principal Investigator — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared with investigators upon reasonable, detailed and written request